CLINICAL TRIAL: NCT03434925
Title: Development of a New Generation Multi Parametric Test for Prediction of Colorectal Neoplasia Recurrence
Brief Title: Multi Parametric Test Predicting the Risk of Colorectal Neoplasia Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Stepan Suchanek, MD., Ph.D., MD., Ph.D., Military University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-31909A
Record Dates: First submitted 2018-01-31; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Colon Cancer
Keywords: colorectal neoplasia; adenoma; colonoscopy; gene mutation; follow-up; recurrence; multiparametric test
MeSH Terms: conditions — Colonic Neoplasms; Adenoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Multi-targeted next generation sequencing — Study directed at finding molecular predictors of recurrent colorectal adenomas also taking into account the intrinsic level of heterogenity imprinted in the internal differences in molecular profiles

SUMMARY:
This project is dedicated to identify the patients with possible higher risk of adenoma recurrence who should have follow-up colonoscopy in yearly interval. As a result, it can lead to optimizing the of follow-up colonoscopies intervals in real-world practice.

DETAILED DESCRIPTION:
In this project, 200 individuals (aged 18 - 75 years) with removed colorectal polyps larger than 10 mm during colonoscopy performed based on all indication (including symptoms and screening procedures) will be included. All procedures will be done with high quality endoscopes (high definition, HD).

In all polyps, the advanced imaging techniques (such as chromoendoscopy and NBI) will be used to determine parts of the polyp suspicious from high-grade dysplasia or cancer. The therapeutic method will be decided by the size and macroscopic appearance of the polyp. In case of flat, sessile polyps and LST lesions (laterally spreading tumors) EMR or ESD will be performed. Pedunculated polyp will be removed by EPE. The goal is to achieve the en-bloc resection. Pathologists (with presence of the endoscopist) will do the first step of histopathology evaluation (cutting the polyp tissue). The aim is to perform the first cut in the most advanced part of the polyp and high density cutting in this area. Standard histopathology evaluation will proceed and will be followed by initial basic molecular testing.

Subsequently, all patients will be observed by colonoscopy in one-year intervals with focus on polyp recurrence. The group of high-risk patients will be selected with at least one of these criteria: 1/ high grade dysplasia adenoma at index colonoscopy; 2/ high score of polyp heterogenity at index colonoscopy; 3/ polyps recurrence at follow-up colonoscopy.

In a high-risk patients group the extensive somatic mutations profiling will be carried out according to multitarget sequencing by NGS technologies (next generation sequencing). Same testing will be done in randomly selected patients not included in the high-risk group, which will be used as a control group for statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal polyp larger than 10mm removed by colonoscopy therapeutic method (EPE, EMR, ESD)
* Signed informed consent with the study and with colonoscopy

Exclusion Criteria:

* FAP, HNPCC and other hereditary CRC syndromes probands
* Recent diagnostic, follow-up or preventive colonoscopy (FOBT-positive colonoscopy, screening colonoscopy) in ≤ 3 years
* Colonoscopy contraindication
* Severe acute inflammatory bowel disease
* Severe comorbidities; likely non-compliance of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of genetic markers for local recurence after resection of colorectal neoplasia | 3 years
  Measurement of gene mutations associated with local recurrence of advanced colorectal neoplasia after endoscopic resection.

SECONDARY OUTCOMES:
Risk of polyp recurrence | 3 years
  Measurement of the number of local recurrences after resection of advanced colorectal neoplasia
Topographic heterogenity of polyps | 3 years
  Measurement of topographical characteristics of colorectal neoplasia (such as demography, histology, tumour genetic heterogeneity and presence of frequently mutated genes) associated with local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Suchanek, MD., Ph.D., Study Director — Military University Hospital
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grega T, Kmochova K, Hejcmanova K, Ngo O, Brodyuk N, Majek O, Bures J, Urbanek P, Zavoral M, Suchanek S. Impact of narrow band imaging in prediction of histology of advanced colorectal neoplasia. Sci Rep. 2025 Jan 9;15(1):1414. doi: 10.1038/s41598-025-85669-w. PMID 39789214